CLINICAL TRIAL: NCT01761799
Title: Protecting Pregnant Women From Infectious Diseases: a Cluster Randomized Evaluation of the Comprehensive "P3" Intervention Package Within Obstetric Practices in Georgia
Brief Title: Protecting Pregnant Women From Infectious Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Saad B. Omer, PhD, Assistant Professor Global Health, Epidemiology, and Pediatrics, Emory University, Schools of Public Health & Medicine & Emory Vaccine Center, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00060292; 5P01TP000300-05 (NIH)
Record Dates: First submitted 2012-12-18; First posted 2013-01-07 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Influenza; Pertussis
Keywords: Influenza; Pertussis; Vaccination
MeSH Terms: conditions — Influenza, Human; Whooping Cough

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- P3 Vaccine Promotion Package (Experimental): The 5 obstetric practices randomized to the intervention arm will receive and implement all components of the evidence-based P3 vaccine promotion package at the beginning of the study.
  Interventions: Behavioral: P3 Vaccine Promotion Package.
- No P3 vaccine promotion package intervention (No Intervention): The 5 obstetric practices randomized to the control arm will not receive the comprehensive vaccine promotion package at the beginning of the study and will instead be instructed to continue their standard of care regarding influenza and Tdap vaccination of pregnant patients.

INTERVENTIONS:
Behavioral: P3 Vaccine Promotion Package. — "P3" stands for Practice, Provider, and Patient level vaccine promotion package. The 5 obstetric practices randomized to the intervention arm will receive this comprehensive influenza and Tdap vaccine promotion package at the beginning of the study. Physicians and staff will be familiarized with each component, and practices will be instructed to implement each component to the best of their ability. The components include: posters, educational brochures, lapel buttons, provider-to-patient talking points, lists of nearby locations offering flu and/or Tdap vaccines (if not offered by the practice), identification of a "vaccine champion" within the practice, provider and staff training on vaccination during pregnancy, and use of an interactive, tablet-based educational tutorial for patients.
  Arms: P3 Vaccine Promotion Package

SUMMARY:
The primary research aim of this project is to test the effectiveness of a comprehensive, evidence-based vaccine promotion package implemented in the obstetric setting on increasing the likelihood that a pregnant woman in Georgia will receive an influenza and/or pertussis vaccine.

DETAILED DESCRIPTION:
The primary research aim of this project is to test the effectiveness of a comprehensive, evidence-based vaccine promotion package implemented in the obstetric setting on increasing the likelihood that a pregnant woman in Georgia will receive an influenza vaccine and/or Tdap vaccine before delivery. A secondary research aim assesses whether the comprehensive package improves maternal knowledge, attitudes, and beliefs regarding maternal and infant vaccination. The intervention package will include evidence-based components aimed at the practice-level, provider-level, and patient level and will be tested through a cluster-randomized trial design. The primary outcome measure is influenza vaccine receipt during pregnancy. The secondary outcomes include 1) receipt of pertussis (Tdap) vaccination during pregnancy, and 2) changes in maternal knowledge, attitudes and beliefs regarding maternal and infant vaccination. The primary hypothesis is that implementation of a comprehensive vaccine promotion package in the obstetric setting will increase the likelihood that a pregnant woman receives an influenza and/or pertussis vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 - 50
* Currently pregnant
* Unvaccinated with 2012 - 2013 seasonal influenza vaccine
* Unvaccinated with Tdap vaccine during current pregnancy

Exclusion Criteria:

* Under 18 years of age or over 50
* Not currently pregnant
* Previous receipt of 2012 - 2013 seasonal influenza vaccine
* Previous receipt of Tdap vaccine during current pregnancy
* Does not speak English

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 330 (Actual)
Dates: Start 2012-12; Primary Completion 2014-02 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Receipt of influenza vaccine during pregnancy | Participants will be followed for the remaining duration of their pregnancy, which will range from approximately 2 weeks to 7 months depending upon their gestation at enrollment.
  Our primary outcome is receipt of a 2012 - 2013 seasonal influenza vaccine during a participant's current pregnancy, before she delivers her child(ren).

SECONDARY OUTCOMES:
Receipt of Tdap vaccine during pregnancy | Participants will be followed for the remaining duration of their pregnancy, which will range from approximately 2 weeks to 7 months depending upon their gestation at enrollment.
  A secondary outcome is receipt of a Tdap vaccine during a participant's current pregnancy, before she delivers her child(ren).

OTHER OUTCOMES:
Changes in maternal knowledge, attitudes and beliefs regarding maternal and infant vaccination | Participants will be followed for the remaining duration of their pregnancy, which will range from approximately 2 weeks to 7 months depending upon their gestation at enrollment.
  This secondary outcome will be assessed through two surveys: one survey administered at baseline upon enrollment, and another survey administered 2 - 3 months post-partum.

CONTACTS AND LOCATIONS:
Overall Officials: Saad B Omer, MBBS,MPH,PhD, Principal Investigator — Emory Unversity
Locations (11):
- United States (11):
  - Athens OBGYN, Athens, Georgia
  - Women's Healthcare Associates, Athens, Georgia
  - Emory Clinic A, Clifton Road Clinic, Atlanta, Georgia
  - Women's Center of Athens, Bogart, Georgia
  - North Pointe OB/GYN, Cumming, Georgia
  - Southern Crescent Women's Health Care, Fayetteville, Georgia
  - W.T. Anderson Health Center - MCCG, Macon, Georgia
  - My OB/GYN, Riverdale, Georgia
  - New Millennium OB/GYN, Riverdale, Georgia
  - Statesboro OB/GYN Specialists, Statesboro, Georgia
  - Shaw Center for Women's Health, Thomasville, Georgia

REFERENCES:
- [Result] Chamberlain AT, Seib K, Ault KA, Rosenberg ES, Frew PM, Cortes M, Whitney EA, Berkelman RL, Orenstein WA, Omer SB. Improving influenza and Tdap vaccination during pregnancy: A cluster-randomized trial of a multi-component antenatal vaccine promotion package in late influenza season. Vaccine. 2015 Jul 9;33(30):3571-9. doi: 10.1016/j.vaccine.2015.05.048. Epub 2015 Jun 1. PMID 26044495
- [Derived] Chamberlain AT, Seib K, Ault KA, Rosenberg ES, Frew PM, Cortes M, Whitney EA, Berkelman RL, Orenstein WA, Omer SB. Impact of a multi-component antenatal vaccine promotion package on improving knowledge, attitudes and beliefs about influenza and Tdap vaccination during pregnancy. Hum Vaccin Immunother. 2016 Aug 2;12(8):2017-2024. doi: 10.1080/21645515.2015.1127489. Epub 2016 Apr 15. PMID 27082036